CLINICAL TRIAL: NCT02155686
Title: Etude de l'Impact Clinique de la télésurveillance à Domicile Par télémédecine de paramètres biométriques de la Personne âgée Polypathologique
Brief Title: Elderly Chronic Diseases Online Biometric Analysis Home Living Technology
Acronym: e-COBAHLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I13027
Record Dates: First submitted 2014-05-24; First posted 2014-06-04 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: The Elderly
Keywords: Elderly; Prevention; Multiple chronic disease; Telemonitoring; Geriatric teleexpertise; Home heath care; Medico-economics
MeSH Terms: interventions — Biosensing Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biosensors (Experimental): Participants in this arm are equipped both with home telecare/automation and with biometric sensors
  Interventions: Device: Biosensors; Device: Home automation
- Automation (Active Comparator): Participants in this arm are equiepd with home automation only
  Interventions: Device: Home automation

INTERVENTIONS:
Device: Biosensors — Device: Biometric sensors; Home automation; telecare
  Arms: Biosensors
Device: Home automation

SUMMARY:
The elderly or people with disabilities want to remain in their homes even when their health condition has been getting worse.

This project aims to demonstrate that home automation and telemonitoring can lead to develop a home safety environment that could help the elderly and individual with disability live independently in their own home.

In this study, the automation sensors containing devices follow up chronic disease clinical factors to monitor their biometrical parameters and detect any abnormal prodromal disease decompensation via telemonitoring and geriatric expertise.

The purpose of this study is:

* to provide clinical evidence of the effectiveness of automation tools and telemonitoring/expertise for the home support for people at risk of loss of autonomy
* to demonstrate the clinical benefit of combining the automation and telemonitoring and geriatric teleexpertise

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 or more.
* House equipped with home automation
* Having been hospitalized in the year prior to the inclusion for the following conditions : heart failure, chronic obstructive pulmonary disease (COPD ), diabetes, high blood pressure ( hypertension ) , repetitive falls, chronic renal failure , stroke, neurodegenerative diseases , malnutrition (according to criteria HAS)
* Multiple chronic diseases (at least 2 comorbidities) .
* Having given free and informed consent

Exclusion Criteria:

* Life expectancy less than 12 months
* Enrolled in another clinical trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 536 (Actual)
Dates: Start 2014-08-27 (Actual); Primary Completion 2018-09-09 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Number of unplanned hospitalization for decompensation | at 12 months
  The effectiveness of home telemonitoring on the cumulative incidence of unplanned hospitalization for decompensation in the elderly

SECONDARY OUTCOMES:
Impact on global health | at 12 months
  * Number of visits to the emergency
  * Number of readmissions
  * Number of days of hospitalization
  * Number of visits to the doctor
Cost/effectivness preventive care | at 12 months
  Evaluate the cost / effectiveness of the impact of telemonitoring on the preventive care in the elderly

CONTACTS AND LOCATIONS:
Overall Officials: Thierry DANTOINE, MD, Study Chair — CHU Limoges
Locations (1):
- Service de Gériatrie - CHU de LImoges, Limoges, France